CLINICAL TRIAL: NCT05307536
Title: Autologous Bone Marrow Mononuclear Cell Transplantation Combined With Educational Intervention for Autism Spectrum Disorders (ASD): A Phase 2 Randomised Controlled Trial
Brief Title: Autologous BMMNCs Combined With Educational Intervention for ASD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISC.19.50
Record Dates: First submitted 2022-02-12; First posted 2022-04-01 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: A total of 54 patients with autism spectrum disorder (3-7 years old) will be recruited and divided into two groups: the controlled group (only intervention education) (n = 27) and the treatment group (Bone marrow mononuclear cell infusions combined educational intervention (n =27)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous BMMNCs infusion combined with educational intervention (Experimental): Bone marrows are harvested from the patient's iliac depending on the patient's body weight as follows: 8 ml/kg for patients under 10 kg; [80 ml + (body weight in kg - 10) × 7 ml] for patients above 10 kg. Mononuclear cells from collected bone marrow are infused intrathecally through a space between number vertebrae 4th and 5th. Two transplantations will be conducted at an interval of 6 months. The educational intervention will be developed based on the Early Start Denver Model for 6 months after the first infusion.
  Evaluation: The efficacy outcomes will be measured using the CARS, Vineland Adaptive Behavior Scales - second Edition (VABS), Autism Behavior Checklists (ABC), and Clinical Global Impression (CGI). In addition, Health-related quality of life (HRQoL) in patients will be evaluated at baseline, two months, six months, and 12 months with those in the control group (educational intervention only) using the Pediatric Quality of Life Inventory (PedsQL)
  Interventions: Combination Product: Autologous BMMNCs transplantation and educational intervention
- Educational intervention (controlled group) (Active Comparator): The educational intervention will be developed based on the Early Start Denver Model for six months after enrollment.
  Evaluation: The efficacy outcomes will be measured using the CARS, Vineland Adaptive Behavior Scales - second Edition (VABS), Autism Behavior Checklists (ABC), and Clinical Global Impression (CGI). In addition, Health-related quality of life (HRQoL) in patients will be evaluated at baseline, two months, six months, and 12 months with those in the control group (educational intervention only) using the Pediatric Quality of Life Inventory (PedsQL)
  Interventions: Combination Product: Educational intervention

INTERVENTIONS:
Combination Product: Autologous BMMNCs transplantation and educational intervention — Biological/ Vaccine: Autologous bone marrow-derived mononuclear cell infusion (BM-MNCs) will be administrated at baseline, and the second infusion will be performed six months after the first administration. For each transplantation, the bone marrow will be harvested through an anterior iliac crest puncture under general anesthesia in the operating theatre. The volume collected depends on the patient's body weight based on our experience from a previous study as follows: 8 ml/kg for patients under 10 kg; [80 ml + (body weight in kg - 10) x 7 ml] for patients above 10 kg but no more than 250 ml in total.
  Educational intervention: 6 months based on the Early Start Denver Model
  Arms: Autologous BMMNCs infusion combined with educational intervention
Combination Product: Educational intervention — Educational intervention: 6 months based on the Early Start Denver Model
  Arms: Educational intervention (controlled group)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of autologous bone marrow mononuclear cell infusion combined with educational intervention for children with autism spectrum disorder (ASD). Inclusion criteria: Male/Female patients diagnosed with Autism disorder based on DSM-V scale, the patient is between 3 to 7 years old, a patient has a medium level to server level of autism (CARS score>=30 to <50), VARS-2 >=50, patient's parent or caregiver must have the educational level of high school or above, patient's family has given consent to participate in the study. Exclusion criteria for treatment group: patient above seven years of age and smaller than 3-year old, autistic patients having epilepsy, hydrocephalus with ventricular drain, allergy to anesthetic agents, severe health conditions such as cancer, failure of heart, lung, liver, or kidney, active infections, children with birth defects of the spine.

DETAILED DESCRIPTION:
A total of 54 patients with autism spectrum disorder (aged 3-7) will be recruited and divided into two groups: the control group (only intervention education) (n = 27) and the treatment group (bone marrow mononuclear cell transplantation combined intervention education (n =27). The bone marrow mononuclear cell will be applied to 27 patients in the treatment group infuse via the intrathecal administration. The primary outcome is measured by the number of AEs/SAEs during BMMNCs infusion. The secondary outcome was measured by clinical examinations performed at baseline and then at 02, 06, and 12 months after the first infusion. Multiple tools were used to diagnose and determine the severity of ASD, including DSM-5, CARS, the Vineland Adaptive Behavior Scales Second Edition (VABS-II), and the Clinical Global Impression (CGI). DSM-5, which was published in May 2013, provides new diagnostic criteria for ASD

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 3 to 7 years old
* Male/Female patient diagnosed with Autism disorder according to the diagnostic criteria for Autism Spectrum Disorder in Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Patient has a medium level to the most severe level of autism (CARS score >=34 to 50)
* Patient's parent or caregiver must have an educational level of high school or above
* Patient's family has given consent to participate in the study

Exclusion Criteria:

* Patient is above seven years of age
* Autistic patient having epilepsy
* Patient with coagulation disorders
* Hydrocephalus with ventricular drain
* Allergy to anesthetic agents
* Sever health conditions such as cancer, failure of heart, lung, liver, or kidney
* Active infections

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2021-12-26 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change of severity of ASD after intervention through the Diagnostic and Statistical Manual of Mental Disorders | 2 months, 6 months, 12 months after the first BMMNCs infusion
  The Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). DSM-5 describes three levels of increasing severity of ASD.DSM-5 describes three levels of increasing severity of ASD, from (1) ("requiring support") to (2) ("requiring substantial support"), and finally to (3) ("requiring very substantial support").
Change of severity of ASD after intervention through the Childhood Autism Rating Scale | 2 months, 6 months, 12 months after the first BMMNCs infusion
  The Childhood Autism Rating Scale (CARS) consists of 14 domains assessing behaviors associated with ASD, with a 15th domain rating general impressions of ASD. Each domain is scored on a scale ranging from one to four; higher scores are associated with a higher level of impairment. Total scores can range from a low of 15 to a high of 60; scores below 30 indicate that the individual is in the non-autistic range, scores between 30 and 36.5 indicate mild to moderate autism, and scores from 37 to 60 indicate severe autism.
Changes in social interaction; adaptive behaviour; daily living skills through Vineland Adaptive Behaviour Scale | 2 months, 6 months, 12 months after the first BMMNCs infusion
  The Vineland Adaptive Behaviour Scale second version (VABS-2) is a semi-structured interview measuring adaptive behavior with standard scores (M = 100, SD = 15). We define proficiency as a standard score of 85 or above (i.e., 1 SD below the mean). This metric for "not impaired" is used in other optimal outcome studies and the learning disability literature. We define growth as an improvement of at least 1 SD in standard scores (15 points) from T1 to T2. Improvement of 1 SD in clinical trials is considered a large effect size.
Changes in social interaction; adaptive behaviour; daily living skills through Clinical Global Impression Improvement | 2 months, 6 months, 12 months after the first BMMNCs infusion
  The Clinical Global Impression Improvement (CGI) is a rating scale that measures symptom severity and treatment response. The severity is categorized into seven levels: 1) not present (no ASD); 2) barely evident ASD symptoms; 3) mild ASD symptoms; 4) moderate ASD symptoms; 5) moderately severe ASD symptoms; 6) severe ASD symptoms or 7) very severe ASD symptoms.
  The response of each patient is also divided into seven levels: level 1) very much improved; level 2) much improved; level 3) minimally improved; level 4) no change; level 5) minimally worse; level 6) much worse; level 7) very much worse.

SECONDARY OUTCOMES:
Changes in health-related quality of life using Pediatric Quality of Life Inventory (PedsQL) | 2 months, 6 months, 12 months after the first BMMNCs infusion
  The Pediatric Quality of Life Inventory™ 4.0 Generic Core Scales - Parent Report (PedsQL) is a tool for assessing the HRQoL of children aged 2-18.
  PedsQL includes four domains (physical functioning, emotional functioning, social functioning, and school functioning) and is scored using three levels: no problems (1), some problems (2), or many problems (3). The PedsQL has 23 items, and scores on the standard portion range from 0 to 100, with 100 representing the best possible quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Liemg Nguyen, PhD, Principal Investigator — Vinmec Research Institute of Stem Cell and Gene Technology
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Vietnam

REFERENCES:
- [Derived] Nguyen LT, Nguyen PM, Nguyen HP, Bui HT, Dao LTM, Van Pham M, Hoang CK, Nguyen PT, Nguyen TTP, Nguyen ATP, Hoang VT, Bui HTP, Vuong NK, Van Ngo D. Outcomes of autologous bone marrow mononuclear cell administration combined with educational intervention in the treatment of autism spectrum disorder: a randomized, open-label, controlled phase II clinical trial. Stem Cell Res Ther. 2025 May 30;16(1):268. doi: 10.1186/s13287-025-04404-4. PMID 40442857
- [Derived] Than UTT, Nguyen LT, Nguyen PH, Nguyen XH, Trinh DP, Hoang DH, Nguyen PAT, Dang VD. Inflammatory mediators drive neuroinflammation in autism spectrum disorder and cerebral palsy. Sci Rep. 2023 Dec 18;13(1):22587. doi: 10.1038/s41598-023-49902-8. PMID 38114596